CLINICAL TRIAL: NCT01500655
Title: Evaluation of Ultrasound-Guided Block of the Lateral Femoral Cutaneous Nerve in Pediatric Patients for Reconstructive Surgical Procedures
Brief Title: Ultrasound-Guided Block of the Lateral Femoral Cutaneous Nerve in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Erik S. Shank, MD, Staff Physician: Pediatric Anesthesiologist, Massachusetts General Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2008P001944
Record Dates: First submitted 2011-12-23; First posted 2011-12-28 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Burns
Keywords: burn; skin graft donor site; analgesia for donor site
MeSH Terms: conditions — Burns | interventions — Catheters

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Catheter (Experimental): An ultrasound guided block of the LFCN is performed, followed by the placement of a catheter underneath the fascia iliaca.
  Interventions: Procedure: Regional nerve block; Procedure: Catheter
- Ultrasound guided LFCN block (Experimental): An ultrasound guided regional nerve block --using ropivacaine 0.2%-- will be performed around the lateral femoral cutaneous nerve (LFCN).
  Interventions: Procedure: Regional nerve block
- Control (No Intervention): This group gets the current standard of care--the donor site is infiltrated with 0.25% bupivacaine.

INTERVENTIONS:
Procedure: Regional nerve block — a block of the lateral femoral cutaneous nerve is performed under ultrasound guidance. For LFCN block, ropivacaine 0.2% will be used. Dose will be 20 ml, unless patient weighs less than 20 kg, in which case volume will be equal to patient's weight in kilograms.
  Arms: Catheter; Ultrasound guided LFCN block
Procedure: Catheter — After an ultrasound guided nerve block is performed a catheter is placed under the fascia iliaca and an infusion of ropivacaine 0.2% running at 0.15 ml/kg/hour is administered for 48 hours.
  Arms: Catheter

SUMMARY:
The purpose of this study is to determine whether either a peripheral nerve block under ultrasound (u/s) guidance of the lateral femoral cutaneous nerve (LFCN), versus an u/s guided block of the nerve followed by continuous catheter infusion of local anesthetic, offers better post-operative analgesia in pediatric burn patients undergoing reconstructive surgery, than the current analgesic regimen of subcutaneous local anesthetic infiltration.

Eligible subject, pediatric patients having reconstructive surgery for burns, having skin graft donor sites of the lateral thighs, will be randomized into three groups: control (having local infiltration of site), ultrasound guided nerve block, or ultrasound guided nerve block with catheter placement --fascia iliac.

Post-operative comfort will be assessed over the next 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* going for reconstructive surgery requiring split thickness skin graft
* patient's donor site will be in distribution of lateral femoral cutaneous nerve
* age >=2 and <22
* patient emotionally/intellectually able to describe intensity of post-op pain using VAS or Wong- Baker faces scale.

Exclusion Criteria:

* potential block/catheter site infected or burned.
* intolerance/allergy to local anesthetics
* BMI > 30
* American Society of Anesthesiologists (ASA) score > 2

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2008-04; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Visual Analog Pain Scale | Q4 hours,while awake, for 48 hours
  We will assess a VAS of pain (0-10)--every 4 hours postoperatively while the patient is awake, for 48 hours post-op.

SECONDARY OUTCOMES:
Narcotic use | 48 hours postoperative
  We will record narcotic requirements of the subjects over the 48 hours post operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Erik S Shank, MD, Principal Investigator — Partners Health Care
Locations (1):
- Shriners Hospital for Children, Boston, Massachusetts, United States